CLINICAL TRIAL: NCT06001645
Title: Pulmonary Interstitial Emphysema (Macklin Effect), Quantitative Imaging Analysis and CytoKine Profiling to Predict Lung Frailty IN ARDS
Brief Title: Laboratory Biomarkers and Pulmonary Interstitial Emphysema in ARDS (PIE-ARDS)
Acronym: PIE-ARDS
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Full Professor, Università Vita-Salute San Raffaele
Other Study IDs: PNRR-MAD-2022-12376
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome; Barotrauma
Keywords: Acute Respiratory Distress Syndrome; Mechanical Ventilation; Intensive Care; Respiratory Failure; Pneumothorax; Macklin effect
MeSH Terms: conditions — Respiratory Distress Syndrome; Barotrauma; Respiratory Insufficiency; Pneumothorax | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and bronchoalveolar lavage fluid will be collected within 12 hours after intubation; blood samples will be centrifuged, and the serum immediately stored at less than 70° C. The following biomarkers will be analysed in the serum and bronchoalveolar lavage fluid: Interleukin-8 (IL-8), Interleukin (IL)-6, IL-1Ra, IL-18, interferon (IFN ), Angiopoietin-2 (Ang-2), Tumour Necrosis Factor receptor-1 (TNFr1), Plasminogen Activator Inhibitor-1(PAI-1), Receptor for Advanced Glycation Endproducts (RAGE), Intercellular adhesion molecule-1 (ICAM-1), Surfactant Protein D (SPD), protein C, Von Willebrand Factor (VWF), CXCL10/CXCR3, and metalloproteases (MMP9, MMP10). Blood and BAL samples obtained from the patients will be placed in specimen tubes (containing heparin for plasma), centrifuged at 1500 G for 10 minutes, and then stored at -70° C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Respiratory Distress Syndrome: Patients with ARDS requiring or not requiring invasive ventilation
  Interventions: Diagnostic Test: Blood and bronchoalveolar fluid collection and analysis; Diagnostic Test: Chest CT scan

INTERVENTIONS:
Diagnostic Test: Blood and bronchoalveolar fluid collection and analysis — Blood and bronchoalveolar lavage fluid will be collected within 12 hours after intubation. Blood samples will be centrifuged, and the serum immediately stored at less than 70° C. The following biomarkers will be analysed in the serum and bronchoalveolar lavage fluid: Interleukin-8 (IL-8), Interleukin (IL)-6, IL-1Ra, IL-18, interferon (IFN ), Angiopoietin-2 (Ang-2), Tumour Necrosis Factor receptor-1 (TNFr1), Plasminogen Activator Inhibitor-1(PAI-1), Receptor for Advanced Glycation Endproducts (RAGE), Intercellular adhesion molecule-1 (ICAM-1), Surfactant Protein D (SPD), protein C, Von Willebrand Factor (VWF), CXCL10/CXCR3, and metalloproteases (MMP9, MMP10). Blood samples obtained from the patients will be placed in specimen tubes containing heparin, centrifuged at 1500 G for 10 minutes, and then the plasma will be aspirated and stored at -70° C. Bronchoalveolar lavage fluid will be centrifuged at 1500 G for 10 minutes to remove cellular contents and stored at -70° C.
Diagnostic Test: Chest CT scan — Computed Tomography Scan per normal clinical practice

SUMMARY:
Barotrauma (pneumothorax, pneumomediastinum) is a well-described complication of Acute Respiratory Distress Syndrome (ARDS), especially in patients with coronavirus disease 2019 (COVID-19) (16.1% in COVID-19, and about 6% in non-COVID-19 ARDS). Macklin effect was recently discovered by our group as an accurate radiological predictor of barotrauma in COVID-19 ARDS; the Investigators also found that density histograms automatically extracted from chest CT images provide a reliable insight into lung composition

. Since lung frailty is a major issue also in non-COVID-19 ARDS, the Investigators want to confirm the predictive role of Macklin effect also in this setting. In addition, the Investigators aim to explore inflammatory profiling to decipher different biological aspects of the same clinical issue. Finally, the Investigators want to develop a specific management algorithm for patients diagnosed, according to our findings, with a specific ARDS sub phenotype characterized by increased lung frailty

DETAILED DESCRIPTION:
Barotrauma occurs frequently in acute respiratory distress syndrome (ARDS), and has a difficult, non-standardized management. Unfortunately, mortality rates remain high (> 60% in COVID-19 ARDS, around 46% in non-COVID-19 ARDS). Interestingly, data from COVID-19 patients suggested that barotrauma may occur also in spontaneously breathing patients with ARDS. Accordingly, frailty of lung parenchyma represents a major issue in ARDS. Protective mechanical ventilation (i.e. ventilation with low tidal volume and low airway pressures) remains a cornerstone of supportive management of ARDS. Unfortunately, mechanical ventilation may worsen pulmonary damage (ventilator-induced lung injury) and, in high-risk patients, may induce barotrauma even when ventilator settings are maintained within the "safe" limit of protective ARDS. Early identification of high-risk features could therefore allow clinicians to individualize management of high-risk patients, by tailoring respiratory support and potentially select candidates for advanced support (i.e. extracorporeal membrane oxygenation) before development of overt barotrauma.

Macklin effect is a well-described radiological sign originally intended to differentiate between "peripheral" (distal airway rupture, "respiratory" barotrauma) and "central" (lesion to large airways/esophaegal injury) causes of air leakage in the mediastinum. However, the Investigators recently identified Macklin effect as a strong radiological predictor of barotrauma development in mechanically ventilated COVID-19 ARDS patients (sensitivity: 89.2%; specificity: 95.6%). In our cohort, radiologically-detected Macklin effect was identified 8-12 days before development of pneumomediastinum/pneumothorax. These preliminary results have been confirmed in a subsequent multicenter study (sample size 697 patients; sensitivity: 100%; specificity: 99.8%).

Furthermore, preliminary data suggest that early application of awake veno/venous extracorporeal membrane oxygenation (ECMO) before invasive mechanical ventilation in COVID-19 patients with severe ARDS and at high-risk for barotrauma (defined as presence of Macklin effect on chest CT imaging) might result in no barotrauma events with a low intubation rate.

Concurrently, a hyper inflammatory sub phenotype has been associated with overall worse outcome both in terms of mortality and ventilator-free days in ARDS. Moreover, the occurrence of lung injury during mechanical ventilation has been proven to be significantly related to the recruitment of mast cells via CXCL10/CXCR3 signaling .

In this view, confirmation of Macklin effect predictive role and identification of further, novel laboratory biomarkers could provide instruments for early risk stratification in ARDS patients.

Taken together, i) quantitative imaging analysis and ii) systemic inflammatory profiling could decipher different biological aspects of the same clinical issue, possibly laying foundation for the definition of a multimodality signature of lung frailty in ARDS patients..

Accordingly, the driving hypotheses of this retrospective/prospective study is that identification of a novel ARDS sub phenotype characterized, irrespective of the underlying etiology, by increased lung frailty could substantially improve the poor prognosis routinely associated with this condition, possibly being a landmark for personalized management strategies.

To further validate the role of Macklin effect, the Investigators will:

* evaluate the accuracy of Macklin effect in a retrospective cohort of 350 ARDS patients (COVID-19 and non-COVID-19)
* identify, throughout densitometry, machine learning and artificial intelligence-based approaches, novel imaging biomarkers characteristics of higher lung frailty in the same cohort.

In the main prospective study, the Investigators will:

* analyse the following biomarkers in the serum and bronchoalveolar lavage fluid of 100 ARDS patients prospectively enrolled: Interleukin-8 (IL-8), Interleukin (IL)-6, IL-1Ra, IL-18, interferon (IFN ), Angiopoietin-2 (Ang-2), Tumour Necrosis Factor receptor-1 (TNFr1), Plasminogen Activator Inhibitor-1(PAI-1), Receptor for Advanced Glycation Endproducts (RAGE), Intercellular adhesion molecule-1 (ICAM-1), Surfactant Protein D (SPD), protein C, Von Willebrand Factor (VWF), CXCL10/CXCR3, and metalloproteases (MMP9, MMP10).
* Develop a specific management algorithm for ARDS patients at high risk for barotrauma by collecting clinical and outcome data from 10 ARDS patients receiving unconventional management (e.g. awake ECMO, ultraprotective ventilation, etc)

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological signs of ARDS, according to Berlin criteria, requiring ICU admission;
* Obtain duly signed informed consent
* Availability of at least one chest CT scan during hospital stay

Exclusion Criteria:

• Poor quality imaging (because of motion/respiratory artefacts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS diagnosis will be enrolled. With the exception of blood and BAL samples collection, all patients enrolled in the prospective cohort will follow their normal course of diagnosis/treatment without any further requirements for the scope of this study other than those provided in the normal management of patients with this condition. Furthermore, any decision regarding drug or procedure will be made by the physician based on her/his clinical judgment, independently from the decision to include the patient in this study. No follow-up medical and/or imaging examinations/laboratory analysis after hospital discharge are needed by the present study design.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically relevant barotrauma | 30 days or until hospital discharge. Specifically, from date of basal CT scan until the date of first radiologically documented barotrauma
  Barotrauma is diagnosed only in the case of clear radiological evidence (free air at chest X-ray and/or chest CT scan).
  Rate of barotrauma will be compared between patients with an hyperinflammatory pattern as compared with control.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - A.O.U. di Cagliari, Cagliari
  - IRCCS San Raffaele Scientific Institute, Milan
  - A.O.U. Pisana, Pisa
  - Ospedale San Carlo, Potenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murayama S, Gibo S. Spontaneous pneumomediastinum and Macklin effect: Overview and appearance on computed tomography. World J Radiol. 2014 Nov 28;6(11):850-4. doi: 10.4329/wjr.v6.i11.850. PMID 25431639
- [Background] Palumbo D, Zangrillo A, Belletti A, Guazzarotti G, Calvi MR, Guzzo F, Pennella R, Monti G, Gritti C, Marmiere M, Rocchi M, Colombo S, Valsecchi D, Scandroglio AM, Dagna L, Rovere-Querini P, Tresoldi M, Landoni G, De Cobelli F; COVID-BioB Study Group. A radiological predictor for pneumomediastinum/pneumothorax in COVID-19 ARDS patients. J Crit Care. 2021 Dec;66:14-19. doi: 10.1016/j.jcrc.2021.07.022. Epub 2021 Aug 12. PMID 34392131
- [Background] Belletti A, Pallanch O, Bonizzoni MA, Guidi L, De Cobelli F, Landoni G, Zangrillo A, De Bonis M, Palumbo D. Clinical use of Macklin-like radiological sign (Macklin effect): A systematic review. Respir Med. 2023 Apr-May;210:107178. doi: 10.1016/j.rmed.2023.107178. Epub 2023 Feb 28. PMID 36863617
- [Background] Paternoster G, Bertini P, Belletti A, Landoni G, Gallotta S, Palumbo D, Isirdi A, Guarracino F. Venovenous Extracorporeal Membrane Oxygenation in Awake Non-Intubated Patients With COVID-19 ARDS at High Risk for Barotrauma. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt B):2975-2982. doi: 10.1053/j.jvca.2022.03.011. Epub 2022 Mar 17. PMID 35537972
- [Background] Maccarrone V, Liou C, D'souza B, Salvatore MM, Leb J, Belletti A, Palumbo D, Landoni G, Capaccione KM. The Macklin effect closely correlates with pneumomediastinum in acutely ill intubated patients with COVID-19 infection. Clin Imaging. 2023 May;97:50-54. doi: 10.1016/j.clinimag.2023.03.003. Epub 2023 Mar 4. PMID 36889115
- [Background] Guarracino F, Baldassarri R, Brizzi G, Isirdi A, Landoni G, Marmiere M, Belletti A. Awake Venovenous Extracorporeal Membrane Oxygenation in the Intensive Care Unit: Challenges and Emerging Concepts. J Cardiothorac Vasc Anesth. 2025 Apr;39(4):1004-1014. doi: 10.1053/j.jvca.2024.12.045. Epub 2025 Jan 9. PMID 39843275
- [Background] Belletti A, D'Andria Ursoleo J, Piazza E, Mongardini E, Paternoster G, Guarracino F, Palumbo D, Monti G, Marmiere M, Calabro MG, Landoni G, Zangrillo A. Extracorporeal membrane oxygenation for prevention of barotrauma in patients with respiratory failure: A scoping review. Artif Organs. 2025 Feb;49(2):183-195. doi: 10.1111/aor.14864. Epub 2024 Sep 21. PMID 39305092